CLINICAL TRIAL: NCT03523819
Title: A Phase Ia/Ib, Open-Label, Dose-Escalation, and Dose-Expansion Study of the Anti-CTLA-4 Monoclonal Antibody CS1002 As Monotherapy and in Combination with Anti-PD-1 Monoclonal Antibody CS1003 in Subjects with Advanced Solid Tumors
Brief Title: A Study of CS1002 in Subjects with Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS1002-101
Record Dates: First submitted 2018-04-22; First posted 2018-05-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-12

CONDITIONS: Solid Tumor, Adult
Keywords: Solid Tumors
MeSH Terms: interventions — Ipilimumab; CS-1003; spartalizumab

STUDY DESIGN:
Masking Description: Randomized for Part 3 of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CS1002 (Experimental): Participants will receive CS1002 intravenously at specified dose on specified days.
  Interventions: Drug: CS1002; Drug: CS1003
- CS1003 (Experimental): Participants will receive CS1003 intravenously at fixed dose on specified days.
  Interventions: Drug: CS1002; Drug: CS1003

INTERVENTIONS:
Drug: CS1002 — Dose levels will be escalated following a modified 3+3 dose escalation scheme
  Other Names: anti-CTLA 4
Drug: CS1003 — Fixed dose at 200mg in combination with CS1002 on a specified dose level
  Other Names: anti-PD1

SUMMARY:
This is a multicenter, open-label, multiple dose, dose escalation phase I study to evaluate the clinical safety, tolerability, PK, and preliminary anti-tumor efficacy of CS1002.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically or cytologically confirmed advanced or metastatic solid tumor(s) for which no effective standard therapy is available or tolerable.
2. ECOG performance status of 0 or 1.
3. Life expectancy ≥12 weeks.
4. Subjects must have adequate organ function
5. Use of effective contraception

Exclusion Criteria:

1. Known brain metastasis or other CNS metastasis that is either symptomatic or untreated.
2. Subjects with active autoimmune diseases or history of autoimmune diseases.
3. Subjects with immunodeficiency or receiving systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to the first dose of CS1002.
4. Has received prior therapy with an anti-CTLA-4 agent.
5. Subjects who had prior chemotherapy, targeted therapy, immunotherapy or any other anti cancer systemic treatment, within 14 days prior to the first dose of CS1002 or who has not recovered from adverse events due to prior therapy.
6. Receipt of major surgical procedure, wide field of radiation, local radiotherapy or radioactive agents within specified time frame prior to the first dose of CS1002.
7. Receipt of live vaccine within 28 days prior to the first dose of CS1002
8. Use of traditional medicinal herbal preparations within 7 days prior to the first dose of CS1002.
9. History of interstitial lung disease or non-infectious pneumonitis except for those induced by radiation therapies.
10. Known history of HIV.
11. Subjects with active Hepatitis B or C infection
12. Subjects with active tuberculosis infection.
13. Subjects with an active infection requiring systemic therapy.
14. History of organ transplantation.
15. History of alcoholism or drugs abuse.
16. History of severe hypersensitivity reactions to other mAbs.
17. Subjects with major cardiovascular diseases.

For more information regarding trial participation, please contact at cstonera@cstonepharma.com

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From the day of first dose to 30 days after last dose of CS1002

CONTACTS AND LOCATIONS:
Overall Officials: Wanmei Wang, Study Director — CStone Pharmaceuticals
Locations (10):
- Australia (8):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Orange Health Service, Orange, New South Wales
  - St Vincent's hospital, Sydney, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Ashford Cancer Centre Research, Adelaide, South Australia
  - Cabrini Health, Malvern, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Boxhill Hospital, Melbourne, Victoria
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No